CLINICAL TRIAL: NCT06272110
Title: Community and NYC Public Healthcare System Partnership to Promote Equitable Access to Language Services and Optimal Preventive Health Services Use Among Individuals With Limited English Proficiency
Brief Title: Promoting Equitable Access to Language Services in Health and Human Services
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 22-01303
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Appropriate Use of Language Across Services
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Post-visit survey of Patients/Caregivers (pre-implementation)
- H+H EHR reports of Patients (pre-implementation)
- Community survey of Community members (pre-implementation)
- Key stakeholder interviews of Patients/Caregivers/Community Members (pre-implementation)
- Key stakeholder interviews of NYC H+H Leadership/Providers/Staff (pre-implementation)
- Key stakeholder interviews of CBO Leadership/Staff (pre-implementation)
- Post-visit survey of Patients/Caregivers (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention
- H+H EHR reports of Patients (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention
- Community survey of Community members (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention
- Key stakeholder interviews of Patients/Caregivers/Community Members (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention
- Key stakeholder interviews of NYC H+H Leadership/Providers/Staff (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention
- Key stakeholder interviews of CBO Leadership/Staff (post-implementation)
  Interventions: Other: System level Language Access (LA) intervention

INTERVENTIONS:
Other: System level Language Access (LA) intervention — Culturally and linguistically appropriate and HL informed strategies and materials/toolkit for community members, patients, and health care providers and staff. Findings from the preparatory work and pre-implementation phase and discussions with key partners will inform the co-design of intervention strategies.
  Groups: Community survey of Community members (post-implementation); H+H EHR reports of Patients (post-implementation); Key stakeholder interviews of CBO Leadership/Staff (post-implementation); Key stakeholder interviews of NYC H+H Leadership/Providers/Staff (post-implementation); Key stakeholder interviews of Patients/Caregivers/Community Members (post-implementation); Post-visit survey of Patients/Caregivers (post-implementation)

SUMMARY:
This is a community-based study that will engage community and health care stakeholders to develop, implement, and evaluate a Health Literacy (HL)-informed, culturally- and linguistically- sensitive approach to improving language access services for patients with limited English proficiency (LEP) to promote health equity and reduce disparities in preventive health services use and health outcomes in New York City (NYC). This study will have a total of 4 phases that include a preparatory work phase (Non-Human Subjects Research), a pre-implementation phase, an implementation phase, and a post-implementation phase.

Findings from the preparatory work and pre-implementation phase and discussions with key partners will inform the co-design of intervention strategies and endpoints for the later phases (implementation and post-implementation phase).

DETAILED DESCRIPTION:
The preparatory work phase (Non-Human Subjects Research) will collect information on policies and procedures related to language access (LA) services use. Educational and patient-facing materials will also be reviewed. This information will be collected pre- and post-implementation.

During the pre-implementation phase surveys and in-depth interviews with key stakeholders will be conducted to assess their views on barriers and facilitators to LA services and preventive services use and ideas about potential intervention strategies and resources to improve these services. Additionally, patients seen for ambulatory care preventive visit at one of the 4 study locations will be invited to complete an anonymous post-visit survey to assess their views on LA services use and provider-patient communication. Community members will also be invited to complete an anonymous survey to assess knowledge of LA rights and satisfaction with LA services. NYC Health & Hospitals (H+H) EHR reports will also be generated to collect visit-level information.

The implementation phase will include the development of culturally and linguistically appropriate and HL informed strategies and materials/toolkit for community members, patients, and health care providers and staff. Findings from the preparatory work and pre-implementation phase and discussions with key partners will inform the co-design of intervention strategies.

During the post-implementation phase surveys and in-depth interviews will be conducted with key stakeholders to assess their views on barriers and facilitators to LA services and preventive services use and ideas about future potential intervention strategies and resources to improve these services. We will also examine perceived appropriateness, acceptability, feasibility, and sustainability of the intervention. We will assess use and adoption of the intervention toolkit. Additionally, patients seen for ambulatory care preventive visit at one of the 4 study locations will be invited to complete an anonymous post-visit survey to assess views on LA services use and provider-patient communication. Community members will be invited to complete an anonymous survey to assess knowledge of LA rights and satisfaction with LA services. H+H EHR reports will also be generated to collect visit-level information.

ELIGIBILITY:
Inclusion Criteria (pre- and post- implementation phase):

Post-visit survey (Patients/Caregivers):

* Patient seen for ambulatory care preventive visit at one of the study locations OR caregiver of a pediatric patient seen for ambulatory preventive visit at one of the study locations.
* 18 years of age and older
* Willingness and ability to participate

H+H EHR Reports:

• Patient seen for ambulatory care preventive visit at one of the study locations

Community survey (Community members):

* Individual that attends community based organizations (CBO) events or uses CBOs' services
* 18 years of age and older
* Willingness and ability to participate

Key Stakeholder interviews:

Patients/Caregivers/Community Members Inclusion Criteria: In order to be eligible to participate, an individual must meet all of the following criteria:

* Prefers to speak in Bengali, French, Spanish, Mandarin, or Polish
* 18 years of age or older
* Patient seen for ambulatory care preventive visit at one of the 4 study locations, caregiver of a pediatric patient seen for ambulatory care preventive visit at one of the 4 study locations OR a community member referred by a CBO
* Willingness and ability to participate

NYC H+H Leadership/Providers/Staff Inclusion Criteria:

* Work at one of the 4 NYC H+H study locations that does language access related work or communicates with patients that prefer to speak a language other than English regularly.
* Leadership (e.g., chief medical officer, Department Director, etc.), provider (Physician, Nurse, Resident), or staff (Interpreter, language access coordinator, clerical staff) at the NYC H+H location
* 18 years of age or older
* Willingness and ability to participate

CBO Leadership/Staff Inclusion Criteria:

* CBO leadership (Director/Coordinator) or staff (Case manager, Patient navigator, etc.)
* 18 years of age or older
* Willingness and ability to participate

Exclusion Criteria (pre- and post- implementation phase):

CBO Leadership/Staff Exclusion Criteria:

* Does not have a working phone number
* Uncorrected hearing impairment

Post-visit survey (Patients/Caregivers):

* Enrolled to key stakeholder interviews
* Does not have a working phone number

H+H EHR Reports (Patients):

• No exclusion criteria

Community survey (Community members):

• Does not have a regular doctor in the US.

Key Stakeholder interviews:

Patients/Caregivers/Community Members Exclusion Criteria:

* Speaks English very well (non-LEP)
* Does not have a working phone number
* Uncorrected hearing impairment

NYC H+H Leadership/Providers/Staff Exclusion Criteria:

* Does not have a working phone number
* Uncorrected hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Post-visit survey: Patients or caregivers of pediatric patients seen for ambulatory care preventive visits. (systematic sampling)
  2. H+H EHR Reports: Patients or caregivers of pediatric patients seen for ambulatory care preventive visits. (systematic sampling)
  3. Community surveys: Individuals that use CBO services or attend their events. (convenience sampling)
  4. Key stakeholder interviews: A purposive variation sample of healthcare staff, CBO staff, patients/caregivers/community members. (purposive sampling)
Sampling Method: Probability Sample
Enrollment: 17500 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of appropriate interpreter use | up to Year 2
Percentage of appropriate interpreter use | up to Year 3

SECONDARY OUTCOMES:
Percentage of patients up to date with preventive screenings and vaccinations | up to Year 2
Percentage of patients up to date with preventive screenings and vaccinations | up to Year 3
Percentage of patients with knowledge of federal rights related to LA services | up to Year 2
Percentage of patients with knowledge of federal rights related to LA services | up to Year 3
Percentage using untrained interpreters | up to Year 2
Percentage using untrained interpreters | up to Year 3
Percentage using recommended HL-informed verbal counseling practices (e.g., teach-back) | up to Year 2
Percentage using recommended HL-informed verbal counseling practices (e.g., teach-back) | up to Year 3
Percentage of patients with satisfaction with LA services preventive health services utilization | up to Year 2
Percentage of patients with satisfaction with LA services preventive health services utilization | up to Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Yin, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Health + Hospitals Diagnostic/Treatment Centers, New York, New York
  - NYC Health + Hospitals/Bellevue, New York, New York
  - NYC Health + Hospitals/Woodhull, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Hsiang.Yin@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Hsiang.Yin@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.